CLINICAL TRIAL: NCT04413201
Title: AFAMOSI: Prospective, Randomized, Multicenter Phase IV Study to Evaluate the Efficacy and Safety of Afatinib Followed by Osimertinib Compared to Osimertinib in Patients with EGFRmutated/T790M Mutation Negative Non-squamous NSCLC in the First-line Setting
Brief Title: AFAMOSI: Efficacy and Safety of Afatinib Followed by Osimertinib Compared to Osimertinib in Patients with EGFRmutated/T790M Mutation Negative Nonsquamous NSCLC
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Hopp (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Michael Hopp, Head of Interdisciplinary Center for Clinical Studies (IZKS), Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFAMOSI; 2019-002197-31 (EudraCT Number)
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Non-squamous NSCLC
MeSH Terms: interventions — Afatinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Afatinib (Experimental): Afatinib followed by osimertinib or ICT depending on T790M status
  Interventions: Drug: Afatinib; Drug: Osimertinib
- Osimertinib (Active Comparator): Osimertinib followed by ICT
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Afatinib — Afatinib followed by osimertinib or ICT
  Other Names: Osimertinib
  Arms: Afatinib
Drug: Osimertinib — Osimertinib followed by ICT

SUMMARY:
This randomized, open label Phase IV trial will be performed in patients with a diagnosis of advanced NSCLC (non-squamous cell histology), harboring EGFR mutation positive but T790M Mutation negative, who have no previous chemotherapy for metastatic NSCLC. Neoadjuvant or adjuvant systemic treatments had to be finished at least (≥) 6 months before study inclusion. In conclusion, this study is investigating the important clinical question whether tumor growth and long term overall survival for a patient is better controlled in a specific treatment sequence of different EGFR-inhibitors. Patients will be treated with registered compounds according to their label in both treatment arms. Thus, all patients will get an effective treatment regimen and patients who progressed on afatinib, and who developed a T790M mutation will be treated subsequently with osimertinib. Those who progressed under osimertinib or under afatinib without T790M mutation will be treated according to the current treatment guidelines with Investigator´s choice of active therapy (ICT) including but not limited to platin doublet chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-squamous NSCLC harboring EGFR mutation positive but T790M mutation negative by local testing
* Unresectable stage UICC ≥ IIIb or metastatic stage UICC IV disease
* TKI naïve for metastatic NSCLC, neoadjuvant or adjuvant chemotherapy allowed
* At least one evaluable lesion according to RECIST v1.1
* Age ≥ 18 years
* ECOG performance status 0 - 2
* Adequate organ function, defined as all of the following:

  1. Absolute neutrophil count (ANC) ≥ 1500/mm3. (ANC > 1000/mm3 may be considered in special circumstances such as benign cyclical neutropenia as judged by the investigator and in discussion with the coordinating investigator)
  2. Platelet count ≥ 75,000/mm3
  3. Estimated glomerular filtration rate (eGFR) > 45 ml/min/1.73 m2 according to the Cockcroft-Gault formula d. If history of cardiac comorbidity: Left ventricular function with resting ejection fraction ≥ 50% or above the institutional lower limit of normal (LLN)

  e. Total Bilirubin ≤ 1.5 times upper limit of normal (ULN), (if related to liver metastases ≤ 3 times ULN). (Patients with Gilbert's syndrome total Bilirubin must be ≤ 4 times institutional upper limit of normal) f. Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤ 3 times the upper limit of normal (ULN) (if related to liver metastases ≤ 5 times ULN)
* Recovered from any previous therapy related toxicity to ≤ Grade 1 at before randomization (except for stable sensory neuropathy ≤ Grade 2 and alopecia)
* Written informed consen

Exclusion Criteria:

* Any investigational drug within 30 days or hormonal anticancer treatment within 2 weeks prior to randomization (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer permitted)
* T790M mutation positive tumors (by local testing)
* Radiotherapy within 2 weeks prior to randomization, except as follows:

  1. Palliative radiation to target organs other than chest may be allowed up to 1 week prior to randomization
  2. Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with coordinating investigator prior to enrolling
* Major surgery within 2 weeks before starting study treatment or scheduled for surgery during the projected course of the study
* Known hypersensitivity to afatinib or osimertinib or the excipients of any of the trial drugs
* History or presence of clinically relevant cardiovascular abnormalities such as

  1. uncontrolled hypertension
  2. congestive heart failure NYHA classification of ≥ 3
  3. unstable angina or poorly controlled arrhythmia as determined by the investigator
  4. Myocardial infarction within 6 months prior to randomization
  5. Clinically important abnormalities in rhythm and conduction as measured by resting electrocardiogram (ECG) (e.g. QTc interval greater than 470 ms) or QTc interval prolongation with signs/symptoms of serious arrhythmia
  6. Congenital long QT syndrome, congestive heart failure, electrolyte abnormalities, or intake of medicinal products that are known to prolong the QTc interval
* Patients with a past or present medical history of

  1. Interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD
  2. Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
  3. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption)
  4. Known active hepatitis B infection (defined as presence of HepB sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier
  5. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 5 years and is considered to be cured
* Pregnancy and contraception:

  1. Women who are pregnant, nursing, or who plan to become pregnant while in the trial
  2. Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at informed consent, for the duration of study participation and for at least 2 months for females and 4 months for males after last dose
* Requiring treatment with any of the prohibited concomitant medications protein Inhibitors/Inductors CYP3A4/5 Inhibitors/Inductors that cannot be stopped for the duration of trial participation or concomitant St. John's Wort
* Uncontrolled brain metastases (Patients with brain or subdural metastases are not eligible, unless they have completed local therapy (≤ 2 weeks apart from last radiotherapy or radiosurgery) and have discontinued the use of corticosteroids, anticonvulsants or have been on stable dose of corticosteroids (i.e. Dexamethasone ≤ 8 mg) for at least 4 weeks before starting study treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before starting study treatment) or Leptomeningeal carcinomatosis 11. Other contraindications to study treatment (Investigators opinion) or legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to EGFR-TKI failure within 24 months for afatinib followed by osimertinib in T790Mpositive group vs osimertinib | 24 months
  The main objective is to investigate whether the time to EGFR-TKI failure at 24 months is better for the treatment sequence of afatinib followed by osimertinib in the T790M positive group compared to osimertinib.

SECONDARY OUTCOMES:
Time to EGFR-TKI failure (afatinib versus osimertinib) | 24 months
  Time from randomization until ICT is indicated
Progression-free survival (PFS: afatinib followed by osimertinib or ICT vs osimertinib followed by ICT) | 24 months
  Time from randomization until disease progression according to RECIST or death
Overall Survival (OS) | 24 months
  Survival Status
Response Rate (RR) | 12 months
  CR+PR according to RECIST
Response Rate (RR) | 24 months
  CR+PR according to RECIST
Disease Control Rate (DCR) | 12 months
  CR+PR+SD according to RECIST
Disease Control Rate (DCR) | 24 months
  CR+PR+SD according to RECIST
Adverse Events | 24 months
  Adverse Events as assessed by intensity of the of the adverse events and the causal relation to trial medication Intensity/Severity: investigator will use the following definitions of severity in accordance with National Cancer Institute common terminology criteria for adverse events, CTCAE, version 5.0; assessment of the relationship of an adverse event to the administration of study drug is a clinical decision by the investigator Institute common terminology criteria for adverse events, CTCAE, version 5.0
Symptom control assessed by patient-reported quality of life (QoL): EQ-5D | 24 months
  patient-reported quality of life assessed by European Quality of Life 5 Dimensions Questionnaire (EQ-5D)
Symptom control assessed by patient-reported quality of life (QoL): EORTC QLQ-C30 | 24 months
  patient-reported quality of life assessed by Questionnaire of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Symptom control assessed by patient-reported quality of life (QoL): EORTC QLQ-LC29 | 24 months
  EORTC QLQ-LC29

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wehler, Prof Dr med, Principal Investigator — Universitätsklinikum Gießen Marburg
Locations (11):
- Germany (11):
  - Klinikum der Ludwig-Maximilians-Universität München, München, Bavaria
  - Universitätsklinikum Gießen Marburg, Giessen, Hesse
  - Sana-Klinikum Offenbach, Offenbach, Hesse
  - Evangelische Lungenklinik Berlin, Berlin
  - Klinikum Bremen-Ost, Bremen
  - Studiengesellschaft Hämato-Onkologie Hamburg, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - Klinikverbund Allgäug gGmbH, Klinik für Pneumologie, c/o Klinik, Immenstadt im Allgäu
  - Gemeinnützige Krankenhausbetriebsgesellschaft Konstanz Mbh, Konstanz
  - Klinik Löwenstein gGmbH, Löwenstein
  - Universitätsklinikum Regensburg, Regensburg